CLINICAL TRIAL: NCT07181993
Title: The Impact of PRISCUS Medication on Fall Risks: A Retrospective Observational Study Based on Medication Data From a Tertiary Hospital
Brief Title: The Impact of PRISCUS Medication on Fall Risks
Status: Active, not recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Daniel Fürstenau, Prof. Dr. rer. pol., Charite University, Berlin, Germany
Other Study IDs: EA2/184/21
Record Dates: First submitted 2025-09-09; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Fall Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Purpose:

This study aims to validate the medication entries in the PRISCUS list-a German expert-based compilation of potentially inappropriate medications for older adults-and to identify additional medications that may pose a fall risk but are not yet included.

Study Design:

This is a retrospective observational study uses electronic health record data from a German research hospital. It includes over 900,000 patient records from multiple departments with a high incidence of falls, covering the period from 2016 to 2022. Statistical analyses, including chi-square tests and propensity score matching, will be employed to evaluate the relationship between medications and fall events.

DETAILED DESCRIPTION:
The PRISCUS list is a catalogue of potentially inappropriate medications for older adults in Germany, derived by experts. However, the validity of its entries has not yet been systematically verified using large-scale patient data. This study aims to validate the current PRISCUS entries and determine whether additional medications should be considered for inclusion based on empirical evidence of an increased risk of falls.

This retrospective study uses data from a German research hospital comprising over 900,000 patient records collected between 2016 and 2022 across 20 clinical departments where falls are common, including oncology, haematology, geriatrics and psychiatry. A total of over 11,000 patients were recorded as having experienced at least one fall event during this period.

Medication data were mapped to German Anatomical Therapeutic Chemical (ATC) codes and linked to clinical records using data from the hospital's pharmaceutical database. Episodes were defined using clinical intervals and various covariates, including age, sex, number of diagnoses and number of procedures, were extracted. Chi-square tests and propensity score matching will be used to compare patients exposed to and unexposed to listed medications, adjusting for key covariates to minimise confounding factors. Candidate medications identified as high risk will undergo further review through clinical evaluation, with additional information sourced from drug package inserts to support risk assessment.

ELIGIBILITY:
Inclusion Criteria:

* All patients across 20 clinical departments with highest fall incidence

Exclusion Criteria:

* Age < 18yrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with patient records between 2016-2022 across 20 clinical departments with highest fall incidence
Sampling Method: Non-Probability Sample
Enrollment: 932912 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Fall Incidents | From January 2016 to October 2022
  In-patients that have experienced a fall within the hospital premises

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Medical Informatics | Charité Universitätsmedizin Berlin, Berlin, State of Berlin, Germany